CLINICAL TRIAL: NCT03330990
Title: A Phase 1 Study to Evaluate the Potential Pharmacokinetic Interaction Between Entrectinib and Midazolam in Cancer Patients
Brief Title: Evaluate the Effect of Entrectinib on the Pharmacokinetics of Midazolam in Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RXDX-101-14; GO40785 (Other: Hoffman-La Roche)
Record Dates: First submitted 2017-10-27; First posted 2017-11-06 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — entrectinib; Midazolam

STUDY DESIGN:
Intervention Model Description: All patients entering this study will receive midazolam and entrectinib.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Entrectinib / Midazolam (Other)
  Interventions: Drug: Entrectinib; Drug: Midazolam Hydrochloride

INTERVENTIONS:
Drug: Entrectinib — 600 mg oral capsule (fasted and fed)
Drug: Midazolam Hydrochloride — 2 mg oral syrup (fasted)

SUMMARY:
This is an open-label study in advanced solid tumor patients to determine if entrectinib affects the pharmacokinetics of midazolam and any of its pharmacologically active metabolites.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria in order to be included in the research study:

1. Histologically or cytologically confirmed diagnosis of advanced or metastatic solid tumors that are not responsive to standard therapies or for which there is no effective therapy.
2. At least 2 weeks or 5 half-lives, whichever is shorter, must have elapsed after prior chemotherapy or small molecule targeted therapy, respectively, at the time of the start of midazolam administration.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status score of ≤1.
4. Adequate hematologic, liver and renal function.
5. Ability to understand the nature of this study and give written informed consent.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from study entry:

1. Participation in another therapeutic clinical trial within 28 days prior to start of midazolam administration.
2. Prior treatment with entrectinib.
3. Known hypersensitivity or intolerance to midazolam or oral formulation excipients, including allergy to cherries.
4. Any condition (in the past 3 months) that may interfere with the conduct of study assessments or may interfere with the interpretation of study results.
5. History of non-pharmacologically induced prolonged QTc interval (e.g., repeated demonstration of a QTc interval > 500 milliseconds from ECGs).
6. Known active infections that may interfere with the conduct of study assessments or may interfere with the interpretation of study results (bacterial, fungal, or viral, including human immunodeficiency virus positive).
7. Other Protocol defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2018-07-11 (Actual)

PRIMARY OUTCOMES:
AUClast | 4 weeks
  Area under the concentration-time curve from 0 to the last measurable concentration of midazolam and the pharmacologically active metabolite 1-hydoxymidazolam in the absence or presence of entrectinib.
AUCinf | 4 weeks
  Area under the concentration-time curve from 0 to infinity of midazolam and the pharmacologically active metabolite 1-hydoxymidazolam in the absence or presence of entrectinib.
Cmax | 4 weeks
  Peak plasma concentration of midazolam and the pharmacologically active metabolite 1-hydoxymidazolam in the absence or presence of entrectinib.
Tmax | 4 weeks
  Time of maximum concentration of midazolam and the pharmacologically active metabolite 1-hydoxymidazolam in the absence or presence of entrectinib.
t1/2 | 4 weeks
  Terminal half-life of midazolam and the pharmacologically active metabolite 1-hydoxymidazolam in the absence or presence of entrectinib.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- United States (3):
  - SCRI-Denver Drug Development Program, Denver, Colorado
  - Florida Cancer Specialists - Sarasota (North Catttlemen Rd), Sarasota, Florida
  - Tennessee Oncology, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No